CLINICAL TRIAL: NCT02573103
Title: Air Pollution and Cardiovascular Disease
Status: Completed | Type: Observational
Sponsor: WeiHuang (Other)
Responsible Party: Sponsor-Investigator, WeiHuang, Peking University School of Public Health, Peking University
Organization: Peking University (Other)
Other Study IDs: WHuang
Record Dates: First submitted 2015-09-28; First posted 2015-10-09 (Estimated); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Metabolic Disorder
MeSH Terms: conditions — Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma and urine
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To determine the effects of ambient airpollution exposures on cardiovascular responses among healthy adults without cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* without CV disease or risk factors (e.g., hypertension, diabetes, or treated hyperlipidemia). Subjects are non-smokers in non-smoking household.

Exclusion Criteria:

* Screening visit BP>140/90 mm Hg, fasting glucose >126 mg/dL, or positive urine pregnancy test (females). Subjects cannot be taking any medications or over-the-counter drugs that affect CV function.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: We will maintain enrollment criteria of the in-progress study being healthy adults without CV disease or risk factors
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2014-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Dyslipidemia | One year
  Analyzed HDL by Beckman AU5800

SECONDARY OUTCOMES:
System oxidative stress | One year
  Analyzed oxidative stress biomarkers,such as MDA by HPLC

CONTACTS AND LOCATIONS:
Overall Officials: Wei Huang, PhD, Principal Investigator — Peking University School of Public Health